CLINICAL TRIAL: NCT04552509
Title: Prospective Evaluation of TRUEBEAM Stereotactic Body Radiotherapy for Localized Prostate Cancer: Risk Stratified MonoTherapy Versus RADIOSURGERY Boost
Brief Title: TRUEBEAM Stereotactic Body Radiotherapy for Localized Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linda Chan, MD (Other)
Responsible Party: Sponsor-Investigator, Linda Chan, MD, Study Principal Investigator, MemorialCare Health System
Organization: MemorialCare Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 790-17
Record Dates: First submitted 2020-09-03; First posted 2020-09-17 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Observation (Other): Observational study of patient efficacy and side effects
  Interventions: Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — Treatment of prostate cancer with stereotactic body radiation therapy (SBRT)

SUMMARY:
The purpose of this study is to determine the effects of TrueBeam stereotactic body radiosurgery in patients with prostate cancer. The device is designed to concentrate large doses of radiation onto the tumor so that injury from radiation to the nearby normal tissue will be minimal. The purpose of this evaluation is to see if this treatment will help patients with your condition and to evaluate the effect of this treatment on your quality of life over time. Radiosurgery is a non-invasive treatment technique used to treat tumors. Despite the word "surgery" in the name, the technology does not remove the tumor with a surgical knife. Instead, a focused, high-intensity beam of radiation targets the tumor, while minimizing dose to surrounding normal healthy tissue.

DETAILED DESCRIPTION:
1.0 BACKGROUND 1.1 Prostatic adenocarcinoma is one of the most common forms of malignancy in men. Every year over 200000 patients are diagnosed with prostate cancer in the United States. Treatment options for these patients include active surveillance, radical prostectomy, external beam radiation therapy, permanent source interstitial brachytherapy and high dose rate (HDR) brachytherapy.

1.2 Each of these treatment options vary in regards to the logistics, anticipated outcomes, and potential side effects of therapy.

1.3 High-dose rate (HDR) brachytherapy has been used in the treatment of prostate cancer since the 1980's with good results. Catheters are placed temporarily in the prostate, and then loaded with a high-dose Iridium-192 source, delivering a few fractions of very high-dose RT. Brachytherapy allows the delivery of conformal, high-dose radiotherapy to the prostate, with a rapid dose fall-off outside of the region. It also takes advantage of low alpha/beta ratio of prostate cancer by using a hypofractionated approach.

1.4 The TrueBeam is a noninvasive radiosurgical system, capable of treating any part of the body from multiple targeting angles, creating a highly conformal three-dimensional radiosurgical treatment volume, guided by orthogonal X-ray-based targeting feedback, and delivering radiation by a highly collimated, robotically controlled linear accelerator. The TrueBeam system targets implanted fiducial markers with sub-millimeter set-up accuracy.

1.5 From a dosimetry standpoint, TrueBeam Stereotactic radiosurgery is capable of producing a dose distribution comparable to that created by prostate HDR brachytherapy treatment, without the need for invasive transperineal catheters, anesthesia, or inpatient admission. It would therefore be possible to deliver the HDR boost portion of a patient's treatment in a non-invasive fashion. As such, the TrueBeam prostate dose fractionation schedule prescribed in this study is based upon prior published prostate HDR brachytherapy experience both as a monotherapy and as a boost to external beam radiation therapy in patients with higher risk disease. The therapeutic volume in this study will also be made to resemble prostate HDR brachytherapy therapeutic volume, with similar dose limitation objectives to the adjacent tissues, including the rectum, bladder and urethra. It is theorized that such an approach should result in similar cancer control rates while lowering overall morbidity and improving the patient's comfort and convenience.

1.6 The feasibility of stereotactic body radiation therapy for treating localized prostate cancer was first described by King at Stanford University. Their phase I protocol delivered 36.25Gy in 5 fractions of 7.25Gy. In a recent report of acute and 18-month late toxicity in 26 "low-risk" patients, no patient experienced grade 3 or 4 acute or late toxicity, and only one patient experienced a grade 2 late morbidity (urethral stricture). Toxicity was less than that reported in MD Anderson's external beam dose escalation trial. Mean PSA 18 months after treatment was 0.22ng/ml. Naples Community Hospital reported a series of more than 70 low and intermediate risk patients treated with the SBRT. The prostate received 35 Gy in 5 fractions of 7 Gy each; acute toxicity was minimal. San Diego Cyberknife, which used a virtual HDR technique, reported a series of more than 124 low and intermediate risk patients treated. The prostate received 38Gy in 4 fractions of 9.5Gy each; acute toxicity was minimal.

1.7 Another potential benefit of stereotactic body radiosurgery relative to HDR brachytherapy is possibly better preservation of potency, even if the radiation distribution is essentially identical between these modalities. This is so because needle trauma has been identified as a potentially significant contributory factor to erectile dysfunction with brachytherapy, including HDR-based monotherapy technique, presumably due to direct physical injury to the neurovascular bundle and/or bulb of the penis, particularly when greater than 13 needle insertions are performed. By comparison, stereotactic body radiosurgery is noninvasive, and so removes this particular erectile dysfunction risk factor.

ELIGIBILITY:
Inclusion Criteria

1. Histologically proven prostate adenocarcinoma

   * Biopsy within 12 months of date of registration required except for patients who already meet criteria for enrollment in the high risk arm of the protocol. For these patients, repeat biopsy will be at the discretion of the treating physician. In general, repeat biopsy is recommended for these patients, but is not required if it will not affect the treating physician's management decisions in regards to the care of the patient.
2. Clinical Stage I-IV, MX-M0 (AJCC 6th Edition)

   * M-stage determined by physical exam, CT, MRI, or Bone Scan. Bone scan not required for Monotherapy Risk Group patients unless clinical findings suggest possible osseous metastases. Bone Scan and contrast CT of the abdomen should be done patients in the Boost Risk Group patients.
3. Prostate volume: ≤ 100 cc (recommended not required)

   * Determined using: volume = π/6 x length x height x width
   * Measurement from CT or ultrasound ≤90 days prior to registration.
4. ECOG performance status 0-1
5. Completion of patient questionnaires in section 4.7.
6. Consent signed

Exclusion Criteria:

1. Prior prostatectomy or cryotherapy of the prostate
2. Prior radiotherapy to the prostate or lower pelvis
3. Implanted hardware or other material that would prohibit appropriate treatment planning or treatment delivery, in the investigator's opinion.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 167 (Estimated)
Dates: Start 2018-06-05 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Local control | 5 years
  Rate of disease recurrence locally

CONTACTS AND LOCATIONS:
Overall Officials: Linda Chan, MD, Principal Investigator — Memorial Health Services
Locations (1):
- MemorialCare Saddleback Medical Center, Laguna Hills, California, United States

IPD SHARING:
Plan to Share IPD: No